CLINICAL TRIAL: NCT04169282
Title: Non-invasive Positive Expiratory Pressure Mask (PEEP-Mask) for Tracheobronchomalacia Associated Cough
Brief Title: PEEP Mask for Tracheobronchomalacia-Induced Cough
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00102498
Record Dates: First submitted 2019-11-14; First posted 2019-11-19 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Tracheobronchomalacia
Keywords: tracheobronchomalacia; TBM; cough
MeSH Terms: conditions — Tracheobronchomalacia; Cough | interventions — Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- nPEP Recipients (Experimental): Single-patient, adjustable expiratory resistance device that provides positive pressure (5 to 20 cm H2O) during expiration
  Interventions: Device: nPEP (non-invasive positive expiratory pressure) mask

INTERVENTIONS:
Device: nPEP (non-invasive positive expiratory pressure) mask — Positive end expiratory pressure (PEEP) mask

SUMMARY:
This study aims to determine if an expiratory resistance device that delivers non-invasive positive expiratory pressure (nPEP) will reduce or stop coughing, reduce airway resistance and improve quality of life in patients with tracheobronchomalacia (TBM) who are not candidates for tracheal stenting.

DETAILED DESCRIPTION:
PROSPECTIVE:

Twenty subjects with chronic cough and TBM diagnosed by bronchoscopy or computed tomography (CT) scan will be recruited to enroll 12 participants. Comorbid conditions that can cause chronic cough, such as asthma, COPD, and GERD, must be treated if present, for subjects to qualify. At the pre-baseline visit (V0), after obtaining verbal informed consent, each subject will complete validated cough questionnaires to quantify their cough severity and cough-related QOL at baseline. The baseline visit (V1) will occur in-person approximately two weeks later, after a run-in period to minimize observation bias related to the cough questionnaires. Written consent will be performed at this visit. At V1, the cough questionnaires will be repeated and subjects' airway resistance and reactance will be measured with impulse oscillometry (IOS). A study physician will perform a physical exam and determine eligibility. Eligible subjects will then be given the nPEP device by the study team and instructed on its use. Approximately four to six weeks after device delivery, at the follow-up visit (V3), cough questionnaires and IOS will be repeated and they will be asked for feedback regarding device design and user experience. Subjects may then be entered into a cohort for up to six additional months, during which there will be no study visits or procedures, but subjects may be contacted by investigators for additional narrative feedback on the device and its use.

Study subjects will be given an nPEP device to use for four to six weeks. During this time participants will be asked to remain on their current medical regimen and not to make any dose changes or add new drugs, unless indicated by their primary care provider. Impulse oscillometry will be measured at V1 and 4-6 weeks later at V3 to assess effect of the nPEP device on airway physiology. A lung CT scan will be performed at V2.

RETROSPECTIVE:

This device was tried on two individuals and it was initiative and was beneficial. Many patients are not candidates for tracheobronchoplasty itself due to medical comorbidities, prefer to avoid the associated risks, or are not candidates for the required tracheal stenting due to trachea size or anatomy. These patients are left without a viable therapeutic option for their severe cough.

Continuous positive airway pressure (CPAP) devices have been reported to stop or prevent cough in TBM, presumably through pneumatic stenting the large airways to maintain their patency during exhalation. CPAP devices, however, are not labeled for this indication and their functional utility is very limited given size of the device, need for a power source, and multiple steps to don the equipment that are not easily completed while actively and uncontrollably coughing.

The physicians aimed to provide positive airway pressure at a low cost and through readily accessible means, in order to abort coughing paroxysms in patients who were not candidates for tracheal stenting and did not have access to commercial CPAP devices. Patients at Duke University Hospital referred to the Interventional Pulmonary service for evaluation of severe, debilitating TBM-related cough and possible tracheal stenting, but who were not candidates for tracheal stenting given their airway anatomy, were given positive end expiratory pressure (PEEP) masks assembled using existing hospital supplies. Specifically, a standard, adjustable (5-20 cm H2O) positive end expiratory pressure (PEEP) valve manufactured for attachment to a manual resuscitation (commonly known as bag-valve-mask) device was attached directly to a flexible face mask, also from a manual resuscitation device. Patients were instructed by their physicians how to use the PEEP masks. The patients used the PEEP mask immediately during their clinical encounter and were given a mask to take home. (The device was created by fellow, Lindsay Boole.)

This was a limited intervention for a very small number of patients (two), specifically identified as being referred to Duke Interventional Pulmonary service with severe cough related to TBM, but with anatomy that ruled them out as candidates for tracheal stenting. There were no formal data collected and no separate follow-up for the purpose of this project (though patients had ongoing clinical follow-up per standard of care). The patients' subjective improvement with the masks was submitted as a case report abstract and poster at the American College of Chest Physician meeting in 2017.

Other physicians asked Dr. Boole about the mask and if it could be used for their patients. Therefore, the investigators would like to request a retrospective review of all patients that used the PEEP mask between January 1, 2009 and August 20, 2019 to be included in this pilot study. Approximately 15 records will be reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Visualization of ≥50% collapse of the trachea or mainstem bronchus on CT scan or bronchoscopy
* No upper or lower respiratory infection within 4 weeks
* Having capacity to provide legal written informed consent

Exclusion Criteria:

* History of tracheobronchoplasty or chronic tracheal stenting
* Current tracheostomy
* History of external chest trauma
* History of:

  * Active treatment for Lung cancer
  * Lung transplantation
  * Unstable congestive heart failure
  * History of spontaneous pneumothorax
* Other medical conditions that interfere with participation in the study
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loretta G Que, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | nPEP Recipients
Started | 10
Completed | 9
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | nPEP Recipients
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Cough Severity as Measured by the Cough Visual Analog Scale (VAS)
Description: The primary objective is to determine if use of the nPEP device will change cough severity. Responses to the Cough VAS range from 0-100 mm, with higher scores corresponding to worse outcomes.
Time Frame: Baseline, two weeks
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | nPEP Recipients
Number analyzed (Participants) | 9
units on a scale | -50.67 (113.00)
Statistical Analysis 1: Comparison: nPEP Recipients; Test type: Superiority; p = 0.108, t-test, 1 sided; paired t-test for normally distributed and transformed data or Wilcoxon's Signed Rank test for non-parametric paired data

2. Primary Outcome: Change in Quality of Life as Measured by the Cough-Specific Quality-of-Life Questionnaire (CQLQ)
Description: The CQLQ score ranges from 28 to 112, with higher scores corresponding to worse outcomes.
Time Frame: Baseline, two weeks
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | nPEP Recipients
Number analyzed (Participants) | 9
score on a scale | -14.63 (10.34)
Statistical Analysis 1: Comparison: nPEP Recipients; Test type: Superiority; p = 0.003, t-test, 1 sided; [statistical method as in outcome 1, analysis 1]

3. Primary Outcome: Change in Quality of Life as Measured by the Leicester Cough Questionnaire (LCQ)
Description: The LCQ score ranges from 19 to 133, with lower scores corresponding to worse outcomes.
Time Frame: Baseline, two weeks
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | nPEP Recipients
Number analyzed (Participants) | 9
score on a scale | 2.53 (3.30)
Statistical Analysis 1: Comparison: nPEP Recipients; Test type: Superiority; p = 0.025, t-test, 1 sided; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Proximal Airway Reactance at 5 Hz (X5) as Assessed by Impulse Oscillometry
Description: The secondary objective is to determine if use of the nPEP device changes airway physiology, specifically proximal airway reactance, as assessed by impulse oscillometry. Reactance at 5 Hz (X5) relates to the physical properties of the lung parenchyma and its ability to expand and facilitate alveolar filling. A more negative X5 value indicates less elasticity of the lung.
Time Frame: Baseline, two weeks
Population: Data not collected on one participant at two weeks.
Measure: Mean (Standard Deviation); unit: cmH2O/L/sec
Arm/Group | nPEP Recipients
Number analyzed (Participants) | 9
cmH2O/L/sec
  Baseline | -3.19 (2.10)
  Two Weeks: number analyzed (Participants) | 8
  Two Weeks | -3.08 (2.37)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | nPEP Recipients
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT04169282/Prot_SAP_001.pdf